CLINICAL TRIAL: NCT05421351
Title: Dynamic Changes in Immune Profile, Neuronal Dysfunction, Metabolomics and Ammonia in Pathogenesis and Therapeutic Response of Hepatic Encephalopathy in Acute-on-Chronic Liver Failure: a Prospective Cohort Study
Brief Title: Immune Profile, Neuronal Dysfunction, Metabolomics and Ammonia in Therapeutic Response of HE in ACLF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, ASSOCIATE PROFESSOR, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: IEC/04/2022-2356
Record Dates: First submitted 2022-05-23; First posted 2022-06-16 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Hepatic Encephalopathy; Acute-On-Chronic Liver Failure; Decompensated Cirrhosis
Keywords: Hepatic Encephalopathy; Acute-On-Chronic Liver Failure; Neurological Dysfunction; Metabolomics; Immune Profiling
MeSH Terms: conditions — Hepatic Encephalopathy; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A total of 8 ml of peripheral blood will be drawn.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experimental: All patients with overt HE in ACLF of any etiology.
- Disease Control Group: 1. Diseased Control patients with Acute-on-Chronic Liver Failure with no Hepatic Encephalopathy
  2. Diseased Control patients with Decompensated Cirrhosis with no Hepatic Encephalopathy
- Control Group 2: Healthy Control without any liver disease

SUMMARY:
There is very little data related to the natural history of disease from covert HE (MHE and grade 1 HE) to overt HE (grades II, III and IV) in ACLF, with implications on long-term neurological recovery after an episode of overt HE. The evolution and pathogenesis of HE is well described in ALF and cirrhosis, but the dynamic changes in HE in ACLF in response to therapy such as ammonia reduction measures, antibiotics to target sepsis and inflammation, measures to alter dysbiosis such as probiotics or fecal microbiota transplant, and measures to target immune dysfunction such as steroids in alcohol-associated hepatitis. The central role of ammonia in the pathogenesis of HE in ACLF has been challenged by recent data. The approach to HE in ACLF has now refocused on systemic and neuro-inflammation, gut dysbiosis, immune dysregulation, and multi-omics approach. Most importantly, the modulation of the metabolome in response to therapy and interventions, and the use of sedatives, paralytic agents, antibiotics etc. in ACLF with HE in a real-world setting has not been reported.

DETAILED DESCRIPTION:
Hepatic Encephalopathy (HE) is a neuropsychiatric disorder characterized by cerebral dysregulation due to hepatic metabolic dysfunction and/or porto-systemic shunting (PSS) resulting in bypass of portal blood flow to the systemic circulation without hepatic detoxification. Hepatic Encephalopathy manifests as a broad spectrum of neurological, cognitive or psychiatric abnormalities ranging from subclinical alterations of cerebral function to coma"(1). Subtle alterations in cerebral function are only detectable by neuropsychological or neurophysiological assessment in minimal hepatic encephalopathy. Weissenborn et al., define HE as a 'significant condition of severe chronic or acute liver insufficiency that is characterized mainly by modifications of motor function, cognition, consciousness, personality. HE was traditionally differentiated into 3 categories as Type A, Type B and Type C. Acute-on-chronic liver (ACLF) has emerged as an independent clinical entity in the field of chronic liver disease which is related to high short-term mortality. The pathogenesis of HE involves blood-derived precipitating factors that cause a neurological deficit in patients with cirrhosis. A major presumption of pathogenesis of HE was assumed to be the central role of ammonia. However, there is now a paradigm shift in our understanding of the etiology, pathogenesis, evolution, and clinical correlation of HE in critically ill patients with cirrhosis and ACLF, wherein systemic inflammation, neuronal dysfunction, cerebral edema, oxidative stress and immune dysregulation are key factors in the multifactorial pathogenesis of HE.

In liver failure, changes in gut microbiota and their by-products like amino acid metabolites, ammonia, endotoxin, oxidative stress, result in neurological transmission alterations like changes in glutamine (Glx), GABA transmission and oxidative stress. Systemic inflammation causes the release of pro inflammatory cytokines such as tumor necrosis factor (TNF)-α, interleukin (IL)-1β and IL-6. They act synergistically with ammonia in developing cognitive dysfunction in patients with HE in and cirrhosis. Currently, there is evidence of the role of neuroinflammation in liver failure. Neuroinflammation is characterized by microglial activation and increased synthesis of the in situ pro-inflammatory cytokines IL-6, IL-1β and TNF-α. Additionally, there is increased gut-liver-brain axis signaling that includes effects of chemokines and cytokines, increased monocytes demand after microglial activation, and changed permeability of the blood-brain barrier(BBB).

However, the exact mechanism by which cerebral edema and HE in ACLF is caused by inflammation is not well known. Thus, identification of novel biomarkers using markers of inflammation, metabolomics, and cerebral imaging techniques to assess the severity of HE in ACLF is essential. The presence of HE is a significant negative predictor of survival in patients with ACLF; hence, studies are needed to fill the gap that is present in the monitoring and prognostication of HE in critically ill patients.

Lactulose is mainstay treatment for HE currently and acts beyond mere ammonia reduction. Lactulose therapy over three months causes a reduction in levels of serum endotoxin, arterial ammonia, inflammatory cytokines and magnetic resonance spectroscopy (MRS) abnormalities(decreased Glx and increased choline and Myo-inositol) (10). Increased cerebral ammonia causes astrocyte swelling and leads to brain edema (11) Hence, most of the drugs used in the HE treatment primarily target ammonia level reduction in the blood. The therapeutic response and progression of HE in ACLF is yet unclear.

ELIGIBILITY:
Inclusion Criteria:

1 . Age 18-65 years 2. Either gender 3. Patients with ACLF (CANONIC definition) of any etiology with HE ≥grade 2 as per West-Haven Criteria

Exclusion Criteria:

1. Patients with structural brain lesions, stroke, diagnosed neurological disease or history of seizures and are on neuropsychiatric medications, like sedatives, antidepressants, or antiepileptic drugs.
2. Severe preexisting cardiopulmonary disease.
3. Patients with hepatocellular carcinoma or systemic malignancy.
4. Post liver transplant patients.
5. HIV/AIDS infection.
6. Patients who are having active COVID-19 infection.
7. Those who do not consent to participate in the study.
8. Those who have TIPS or Porto systemic surgical shunt in situ.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Experimental group (A1) n=75 Disease Control Group (A2) [ACLF without HE (n=20)], [Decompensated Cirrhosis without HE (n=20)] Healthy Control group-20
Sampling Method: Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2022-10-02 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Baseline Assessment of dynamic markers of systemic inflammation (IL-1, IL-6, TNF alpha, CD163, CD10, etc) following HE specific management strategies in ACLF. | Day 0
  Systemic inflammation and Immune profiling will be accessed by Flow Cytometry
Changes in markers of systemic inflammation (IL-1, IL-6, TNF alpha, CD163, CD10, etc) following HE specific management strategies in ACLF. | Day 7
  Systemic inflammation and Immune profiling will be accessed by Flow Cytometry
MR Imaging of HE in ACLF | MRI-MRS (At time of Discharge from Hospital)
  MRI-MRS
Assessment of markers of neuronal dysfunction in HE in ACLF | Day 0
  Neuronal dysfunction markers will be assessed by ELISA for GFAP, S110B, etc
Change in markers of neuronal dysfunction in HE in ACLF | Day 7
  Neuronal dysfunction markers will be assessed by ELISA for GFAP, S110B, etc
Assessment of conventional markers of HE and clinical outcomes using standard tests like arterial ammonia, WHC and CHESS scores and severity scores of ACLF like (CLIF-C-ACLF/MELD Na). | Day 0
  Ammonia will be assessed by PocketChem BA Blood Ammonia meter. WHC, CHESS will be assessed for encephalopathy and severity score will be calculated using blood investigation.
Assessment of conventional markers of HE and clinical outcomes using standard tests like arterial ammonia, WHC and CHESS scores and severity scores of ACLF like (CLIF-C-ACLF/MELD Na). | Day 4
  Ammonia will be assessed by PocketChem BA Blood Ammonia meter. WHC, CHESS will be assessed for encephalopathy and severity score will be calculated using blood investigation.
Assessment of conventional markers of HE and clinical outcomes using standard tests like arterial ammonia, WHC and CHESS scores and severity scores of ACLF like (CLIF-C-ACLF/MELD Na). | Day 7
  Ammonia will be assessed by PocketChem BA Blood Ammonia meter. WHC, CHESS will be assessed for encephalopathy and severity score will be calculated using blood investigation.
Baseline Metabolomics in patients with HE in ACLF | Day 0
  Metabolomics will be performed by LC/GC-MS to find putative metabolites associated with HE
Change in Metabolomics following specific management strategies for HE in ACLF and standard medical management of ACLF. | Day 7
  Metabolomics will be performed by LC/GC-MS to find putative metabolites associated with HE

SECONDARY OUTCOMES:
Predictors of HE resolution in ACLF | Day 90
  Predictability for outcomes of HE resolution and survival will be compared between novel biomarker and conventional tests
New hospitalization till 90 days after enrolment. | Day 90
  Patient will be followed for 90 days to assess re-hospitalization and recurrence of HE

CONTACTS AND LOCATIONS:
Overall Officials: Dr Madhumita Premkumar, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No